CLINICAL TRIAL: NCT05511805
Title: Investigation of the Relationship Between Pain, and Balance, Proprioception in the Knee, the Strength of the Erector Spinae and Multifidus Muscles in Individuals With Non-Specific Low Back Pain
Brief Title: Examination of Pain in Individuals With Non-Specific Lack Pain
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: 12/37
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2022-09

CONDITIONS: Back Pain; Balance; Proprioception
Keywords: Low back pain; Balance; Proprioception
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Visual Analogue Scale (VAS), — The pain levels of the individuals participating in the study will be evaluated with the Visual Analog Scale. According to VAS, in the severity of pain; '0' means no pain, '10' means worst pain imaginable. During the study, the participants will be asked to rate their pain experienced in daily life and pain during evaluation between 0-10 points. Individuals with pain intensity of 3 and above according to VAS will be included in the study.
Other: Oswestry Low Back Pain and Disability Questionnaire — The Oswestry scale will be used to determine the level of functional disability due to low back pain. In this questionnaire, 10 questions are asked about pain intensity, social life, weight lifting, walking, personal care, sitting, sleeping, sexual life, standing and travel. Each question has 6 options and the patient is asked to choose the statement that best describes his or her condition.
Other: Functional Low Back Pain Scale — The Functional Low Back Pain Scale will be used to evaluate how much the low back pain experienced by the people who will be included in the study affects their daily living activities. Evaluated functions; work and school activities, home activities, wearing shoes or socks, leaning forward, lifting an object from the ground, habits, sleeping, walking, sitting, climbing stairs, standing and driving. The questionnaire consists of 12 questions, and each item scores in the range of 0-5 points.
Device: Prokin TecnoBody isokinetic balance 2 device — For the one-leg balance test, the subject is positioned on one leg at the origin of the platform. The participant is asked to look at any stationary point or object in front of him. Participants are allowed to experiment on the platform of the meter for approximately 2-3 minutes. The stem sensor apparatus is then attached to coincide with the xiphoid projection. After the torso sensor is attached, the patient is placed in the dominant side position on one foot and the static balance test measurement is started. 30 seconds from the patient in this position. asked to stop.
Device: EMG — In our study, electromyography (EMG) device will be used to evaluate muscle strength. Electromyography is a method by which electrical activity analysis of muscles can be performed. In the study, the erector spina and multifidus muscles will be measured. Measurements are made with electrodes placed on the skin surface.
Device: Algometer — The pressure perception and pain threshold of pain sensitivity are determined and recorded with an algometer. The details of the application will be explained to the participant and it will be emphasized that the feeling of pressure he feels causes pain and that he should give a 'stop' command. The pressure force is increased until the patient receives the 'stop' command in the area to be applied. It is stopped by the command from the patient and the response on the algometer screen is recorded. These measurements are repeated 3 times. The average of these three recorded measurements is determined.
Device: Goniometer — Using the universal goniometer's measure of knee joint range of motion, sense of proprioception will be evaluated. For measurement, subjects are asked to lie on a stretcher in the prone position. The pivot point of the goniometer is placed in the center of the lateral knee joint condyle. The fixed arm of the goniometer is fixed in parallel at the level of the thoracantary major, and the movable arm is positioned at the level of the head of the fibula and the lateral malleolus. First of all, starting from the 0° extension position to the knee joint, the angle desired by the physiotherapist is made and the value in the goniometer is recorded. Then, the patient is asked to bring the knee joint, which is still in 0° extension, to the angle brought by the physiotherapist. Then the angle brought by the patient to the knee joint is recorded.

SUMMARY:
The aim of this study is to examine the relationship between pain, and balance, proprioception sensation in the knee, erector spinae and multifidus muscle strength in individuals with non-specific low back pain.

DETAILED DESCRIPTION:
Impaired postural control in people with non-specific low back pain; It can be affected by many factors such as pain, musculoskeletal disorders, proprioception. Postural control is important for the continuation of activities of daily living. Postural control is decreased in patients with non-specific low back pain. According to the proprioception examinations, patients with low back pain are more impaired than healthy individuals. Impaired proprioception can also reduce the ability to maintain posture, balance control and increase the load on the spine. Thus, individuals with low back pain may become more vulnerable to injuries. Weakness of the abdominal muscles and superficial trunk muscles are also risk factors for low back pain.

Weakness and fatigue may occur as a result of structural changes, which are more common in the paraspinal muscles and the multifidus muscle. This can lead to deterioration of lumbar stability. Because these muscles have an important place in providing stability.

Proprioceptive information from the hip, knee and ankle and coordination of the joints are important in maintaining and controlling balance. Regional receptors in muscles, joints, skin and tendons and proprioception in the knee joint provide the necessary joint activity and stabilization. With the decrease in balance and proprioception, pain may occur, and we may encounter a decrease in muscle strength as a result of leading a sedentary life. In this case, since the proper posture, muscle activity and balance required for coordinated movement are negatively affected, the movement is impaired. Because these activities must be performed in the correct order for the movement to occur.

In the literature, there are studies on the relationship of low back pain with muscle strength, balance and proprioception; however, the lack of sufficient studies investigating the relationship between balance and proprioception in the knee in individuals with non-specific low back pain suggests that the study to be conducted will make an important contribution to the literature and reveals the importance of our study.

ELIGIBILITY:
Inclusion Criteria:

* Having pain intensity of 3 or more according to VAS.
* Having a mini mental test score of 24 and above
* Being able to stand on one leg.
* Having low back pain for 3 months or more

Exclusion Criteria:

* Osteoporosis
* Being in the 0%-20% range on the Oswestry scale
* Pregnancy
* Being on constant painkillers for one reason or another
* Having undergone lumbar, hip, knee and ankle surgery.
* Having severe hearing, vision, speech impairment

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with non-specific low back pain.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain | Baseline
  This was evaluated using the Visual Analogue Scale (VAS). According to VAS, in the severity of pain; Generally, '0' means no pain, and '10' means the worst pain imaginable.
Evaluation of static stance on one leg | Baseline
  This was evaluated with Prokin TecnoBody isokinetic balance 2 device. After the torso sensor was attached, the patient was placed in the dominant side position on one foot and the static balance test measurement was started. The patient is expected to stand in this position for 30 seconds.The test was started by pressing the start button on the computer keyboard connected to the device. The test was automatically terminated by the computer when it expired. A computer printout containing the static test evaluation results was obtained.
Evaluation of back extensor strengths | Baseline
  These were evaluated with EMG. In the study, measurement of erector spina and multifidus muscles was performed. Measurements were performed with electrodes placed on the skin surface to measure the total activity of the muscles and to determine muscle fatigue non-invasively.
Evaluation of low back pain thresholds | Baseline
  This was evaluated with Algometer. Determination of pressure perception and pain threshold of sensitivity to pain was determined and recorded with an algometer. It was standardized to perform the measurements on the determined -region-. The details of the application were explained to the participant, and it was emphasized that the pressure sensation he felt caused pain and that he needed to give a 'stop' command. It was stopped with the command received from the patient and the response on the algometer screen was recorded.
Evaluation of the effect of pain on functionality | Baseline
  It is a scale used to evaluate the extent to which low back pain experienced by patients affects their functions in daily life. Evaluated functions; work and school activities, home activities, wearing shoes or socks, bending forward, lifting an object from the ground, habits, sleeping, walking, sitting, climbing stairs, standing and driving. This questionnaire consists of 12 questions. Each item has a score in the range of 0 - 5 points. The minimum possible score is "0", and the maximum possible score is "60". 60 points; states that the activities in the questionnaire were not difficult.
Evaluation of the level of functional disability | Baseline
  It is a scale used to determine the level of functional disability due to low back pain. This scale consists of ten questions. Each question has a score between zero and five. In this questionnaire, the severity of pain, social life, lifting, walking, personal care, sitting, sleeping, standing, traveling, the level of pain and the degree of change in pain are questioned.
Evaluation of the proprioception | Baseline
  The sense of proprioception was evaluated by using the joint range of motion measurement of the universal goniometer. The subjects were asked to lie on the stretcher in the prone position to measure the range of motion of the knee joint. The pivot point of the goniometer was determined as the lateral knee joint condyle and placed. The fixed arm of the goniometer was fixed in parallel at the level of the trochanter major, and the movable arm was positioned at the level of the head of the fibula and the lateral malleolus. First of all, the knee joint is started from 0° extension position and brought to the angle desired by the physiotherapist and the value in the goniometer is recorded. Then, the patient is asked to bring the knee joint, which is again in 0° extension, to the angle brought by the physiotherapist. By following the knee joint flexion of the movable arm, the angle that the patient brings the knee joint is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Pehlivan, Assoc. Prof., Study Director — Saglik Bilimleri University
Locations (1):
- Sağlık Bilimleri Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nowotny AH, Calderon MG, Alves BMO, de Oliveira MR, Andraus RAC, Aguiar AF, Amorim CF, Leonard G, da Silva RA. Low-Back Pain and Knee Position-Related Differences on Postural Control Measures During a One-Legged Stance in Athletes. J Sport Rehabil. 2020 Nov 25;30(4):631-637. doi: 10.1123/jsr.2020-0095. PMID 33238243
- [Background] Goubert D, Oosterwijck JV, Meeus M, Danneels L. Structural Changes of Lumbar Muscles in Non-specific Low Back Pain: A Systematic Review. Pain Physician. 2016 Sep-Oct;19(7):E985-E1000. PMID 27676689
- [Background] Ruhe A, Fejer R, Walker B. Is there a relationship between pain intensity and postural sway in patients with non-specific low back pain? BMC Musculoskelet Disord. 2011 Jul 15;12:162. doi: 10.1186/1471-2474-12-162. PMID 21762484
- [Background] Hlaing SS, Puntumetakul R, Wanpen S, Boucaut R. Balance Control in Patients with Subacute Non-Specific Low Back Pain, with and without Lumbar Instability: A Cross-Sectional Study. J Pain Res. 2020 Apr 23;13:795-803. doi: 10.2147/JPR.S232080. eCollection 2020. PMID 32425585
- [Background] Hodges P, van den Hoorn W, Dawson A, Cholewicki J. Changes in the mechanical properties of the trunk in low back pain may be associated with recurrence. J Biomech. 2009 Jan 5;42(1):61-6. doi: 10.1016/j.jbiomech.2008.10.001. Epub 2008 Dec 4. PMID 19062020